CLINICAL TRIAL: NCT06366594
Title: Effectiveness of First-line Nurse Manager Authentic Leadership Training Program on Nurses' Attitudes in Medical and Surgical Care Units
Brief Title: First-line Nurse Manager Authentic Leadership Training Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matrouh University (Other)
Responsible Party: Principal Investigator, Nagah Abd El-Fattah Mohamed Aly, Assistant professor of Nursing administration, Matrouh University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 0305897
Record Dates: First submitted 2024-04-03; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Intervention
Keywords: leadership; Training program; Nurse manager; Nurse; Self-efficacy; Trust

STUDY DESIGN:
Intervention Model Description: A quasi-experimental research design
Who Masked: Participant
Masking Description: A quasi-experimental design utilized one group for pre-, post, and follow-up intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of first-line nurse managers (Other): First-line nurse managers received an authentic leadership training program
  Interventions: Behavioral: Authentic leadership training program
- Intervention Group (Other): First-line nurse managers received an authentic leadership training program
  Interventions: Behavioral: Authentic leadership training program

INTERVENTIONS:
Behavioral: Authentic leadership training program — 37 first-line nurse managers received authentic leadership training program

SUMMARY:
Authentic leadership behavior is considered a mandatory strategy for enhancing the nurse manager capabilities and practice as well as achieving positive nurses' attitudes.

DETAILED DESCRIPTION:
Authentic leadership behavior is considered a mandatory strategy for enhancing the nurse manager's capabilities and practice as well as achieving positive nurses' attitudes. This study aimed to investigate the effectiveness of authentic leadership programs for first-line nurse managers on nurses' attitudes, including nursing care self-efficacy and trust.

ELIGIBILITY:
Inclusion Criteria:

First-line nurse managers

* willing to participate in the study
* work in medical and surgical wards
* Sign a consent

Exclusion Criteria:

* First-line nurse managers

  * work in outpatient units and other wards
  * Did not sign a consent
  * Absent from training

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Questionnaire to measure first-line nurse managers' knowledge about authentic leadership | one month
  Fist-line nurse managers' knowledge about authentic leadership as assessed using dichotomous scale (No =0, Yes=1). Change in nurse managers' knowledge level in one month
questionnaire to measure authentic leadership behavior among first-line nurse managers | one month
  Fist-line nurse managers' authentic leadership behavior as assessed using five-point Likert scale. Change in nurse managers' behavior level in one month
Questionnaire to measure nursing care self-efficacy | one month
  nursing care self-efficacy was assessed using a 10-point Likert scale (0 =cannot do at all) to 10=certainly can do) perceived self-efficacy as assessed using a 10-point Likert scale (0 =cannot do at all) to 10=certainly can do).
Questionnaire to measure nurses' trust in their workplace | one month
  Nurses' trust in their workplace as assessed using a five point Likert scale (1 =strongly disagree to 5=strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Nagah Abd El-Fattah Mohamed Aly, Ph.D, Principal Investigator — Faculty of Nursing, Matrouh University, Egypt; Wael M. Lotfy, Ph.D, Study Director — Faculty of Nursing, Matrouh University, Egypt; Safaa M. El-Shanawany, Ph.D, Study Chair — Forensic Medicine and Clinical Toxicology, Faculty of Medicine, Alexandria University, Egypt; Maha Ghanem, Ph.D, Study Chair — Forensic Medicine and Clinical Toxicology, Faculty of Medicine, Alexandria University, Egypt; Hanaa Abbass, Ph.D, Principal Investigator — Faculty of Nursing, Matrouh University , Egypt
Locations (1):
- Faculty of Nursing, Matrouh University, Marsá Maţrūḩ, Egypt

IPD SHARING:
Plan to Share IPD: No